CLINICAL TRIAL: NCT06843083
Title: Contrast-Enhanced Mammography or Breast MRI: Which Choice for Optimal Diagnostic Performance?
Brief Title: Contrast Enhanced Mammography or Breast Magnetic Resonance: Which Choice for Optimal Diagnostic Performance?
Acronym: CEM MRI choice
Status: Enrolling by invitation | Type: Observational
Sponsor: Graziella di Grezia (Other)
Collaborators: Link Campus University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Graziella di Grezia, principal investigator, Link Campus University
Organization: Link Campus University (Other)
Other Study IDs: T_2_2025
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Prevention; Breast Cancer Diagnosis
Keywords: contrast enhanced mammography; breast MRI; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CEM Group: CEM Group:
  Patients in this group will undergo Contrast-Enhanced Mammography (CEM) as part of their diagnostic imaging workup for breast lesions. The CEM procedure will be used to evaluate the sensitivity and specificity of this imaging technique in detecting and characterizing breast lesions in patients with dense breast tissue or inconclusive findings from standard mammography.
  Interventions: Diagnostic Test: CEM protocol
- MRI Group: MRI Group:
  Patients in this group will undergo Breast Magnetic Resonance Imaging (MRI), which will be used to evaluate the diagnostic accuracy of MRI in detecting and characterizing breast lesions. The MRI procedure will be compared with CEM to assess the differences in diagnostic performance, sensitivity, specificity, and clinical impact in managing patients with high-risk factors or dense breast tissue.
  Interventions: Diagnostic Test: breast MRI

INTERVENTIONS:
Diagnostic Test: CEM protocol — CEM combines low-energy mammography with high-energy contrast-enhanced imaging to highlight areas of neo-angiogenesis, which are indicative of malignancy. This intervention will be used to evaluate the diagnostic performance of CEM in detecting and characterizing breast lesions, especially in patients with dense breast tissue or inconclusive findings from routine mammography.
  Other Names: CEM
  Groups: CEM Group
Diagnostic Test: breast MRI — MRI (Magnetic Resonance Imaging):
  MRI will be used as an alternative imaging modality for breast lesion detection and characterization. MRI provides detailed soft tissue imaging and is widely used in the evaluation of high-risk patients or those with dense breast tissue. The results from MRI will be compared to CEM findings to determine which modality offers superior diagnostic accuracy and clinical impact.
  Groups: MRI Group

SUMMARY:
This study compares the diagnostic performance of Contrast-Enhanced Mammography (CEM) and Breast MRI in evaluating breast lesions. It aims to assess sensitivity, specificity, and diagnostic accuracy to identify the optimal imaging modality for clinical scenarios such as dense breast tissue and high-risk populations.

DETAILED DESCRIPTION:
Search differences and performance of MRI and CEM

ELIGIBILITY:
Inclusion Criteria:

* Age: Women aged 18 years and older.
* Indication for Advanced Imaging: Patients referred for Contrast-Enhanced Mammography (CEM) or Breast MRI due to suspicious findings or high-risk factors for breast cancer.
* Dense Breast Tissue or Inconclusive Findings: Patients with dense breast tissue or inconclusive results from standard mammography.

Informed Consent: Ability to provide written informed consent for participation in the study.

- Presence of Breast Tissue: Female or transgender women who have breast tissue suitable for imaging.

Exclusion Criteria:

* Contraindications to MRI: Patients with contraindications to Breast MRI (e.g., implanted pacemakers, severe claustrophobia, or metallic implants that cannot be removed).
* Contraindications to Contrast Agents: Patients who have allergies or contraindications to iodinated contrast agents used in CEM.

Severe Renal Impairment: Patients with severe renal impairment (eGFR < 30 mL/min/1.73 m²), as they may not safely undergo contrast-enhanced imaging.

* Pregnancy or Breastfeeding: Women who are pregnant or breastfeeding, as the use of contrast agents may pose risks to the fetus or infant.
* Already Confirmed Primary Tumor: Patients with a confirmed primary breast malignancy or another primary tumor site (e.g., gastrointestinal, lung) that has already been diagnosed.
* Other Medical Conditions: Patients with serious medical conditions that may interfere with participation in the study or may affect the safety of the imaging procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult women aged 18 years or older who are referred for advanced breast imaging due to suspicious breast lesions or high-risk factors for breast cancer. The population will include individuals with dense breast tissue or those who have had inconclusive findings from standard mammography, making them candidates for Contrast-Enhanced Mammography (CEM) or Breast Magnetic Resonance Imaging (MRI).
  The study aims to include a diverse cohort of patients, both in terms of age and background, as long as they meet the inclusion criteria and do not fall under the exclusion criteria. The study will be conducted at ASL Avellino, Italy, and will involve patients from various risk groups, including those with a family history of breast cancer, personal history of other cancers, and those with dense breast tissue who may require advanced imaging for accurate diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of CEM vs. MRI for Breast Lesion Detection and Characterization | From enrollment to the end of treatment at 12 months
  The primary outcome of the study is to compare the diagnostic accuracy of Contrast-Enhanced Mammography (CEM) and Breast Magnetic Resonance Imaging (MRI) in detecting and characterizing breast lesions. This will be assessed by evaluating the sensitivity, specificity, and overall diagnostic performance of both imaging modalities. Findings will be correlated with histopathological results or follow-up imaging to determine the accuracy of each modality in the diagnosis of breast cancer.

SECONDARY OUTCOMES:
Sensitivity and Specificity of CEM vs. MRI | From enrollment to the end of treatment at 12 months
  This secondary outcome aims to compare the sensitivity and specificity of CEM and MRI in detecting breast lesions. Sensitivity refers to the ability to correctly identify true positives, while specificity refers to correctly identifying true negatives. These metrics will be analyzed to assess the diagnostic capability of each imaging technique.
Positive Predictive Value (PPV) and Negative Predictive Value (NPV) of CEM vs. MRI | From enrollment to the end of treatment at 12 months
  The positive predictive value (PPV) and negative predictive value (NPV) will be calculated for both CEM and MRI. PPV indicates the proportion of positive test results that are true positives, while NPV indicates the proportion of negative test results that are true negatives.
Patient Preference and Tolerability of CEM vs. MRI | From enrollment to the end of treatment at 12 months
  This outcome will assess patient preference and tolerability between CEM and MRI. Patients will be asked to complete a questionnaire regarding their comfort during each imaging procedure, and their preference for one modality over the other will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No